CLINICAL TRIAL: NCT02972229
Title: Whole Versus Partial Vertebral Body IMRT for Spinal Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhenwei Zou, Principal Investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WuhanUH201610
Record Dates: First submitted 2016-11-16; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- partial body group (Experimental): 10x(3-5) Gy IMRT on partial vertebral body
  Interventions: Radiation: 10x(3-5) Gy IMRT
- whole body group (Active Comparator): 10x3 Gy IMRT on whole vertebral body
  Interventions: Radiation: 10x3 Gy IMRT

INTERVENTIONS:
Radiation: 10x(3-5) Gy IMRT — 10x(3-5) Gy IMRT on partial vertebral body for spinal metastases
  Arms: partial body group
Radiation: 10x3 Gy IMRT — 10x3 Gy IMRT on whole vertebral body for spinal metastases
  Arms: whole body group

SUMMARY:
To compare the treatment effect and toxicity between Intensity-Modulated Radiation therapy for whole metastatic vertebral body and simple metastatic lesions of vertebra in metastatic spinal tumors

DETAILED DESCRIPTION:
This study is a prospective, randomized, single center, controlled explorative study in the parallel-group design to evaluate the difference in clinical outcomes for patients with metastatic spine disease treated with a whole versus partial vertebral body contouring approach. Thereby two different techniques were evaluated: whole vertebral body (WB) group with 10 x 3Gy or partial vertebral body (PB) group with 10x (3-5)Gy. Prior to their enrolment into the study, the patients will undergo a staging of the vertebral column in connection with their radiation-planning computed tomography (CT) and MRI to measure the myelon dimension. After the baseline results have been recorded, the patients will be randomized into one of the two groups: PB group RT 10x (3-5) Gy (n = 30) or WB group RT 10 x 3 Gy (n = 30). The target parameters will be measured and recorded at baseline, at 1 to 2 weeks; and at months 2 to 3, 4 to 6 and 7 to 12 after treatment.

The primary endpoint was the time to pain relief. Secondary endpoints were quality of life (QoL), fatigue, pain, overall survival, bone survival, local control, pathological fracture, pain-free internal and neurological deficit. The baseline examination shall be carried out on the first day of radiotherapy prior to the start of therapy and is scheduled to comprise the comprehensive recording of the sociodemographic data, the recording of the current pain situation, the quality of life, and the current degree of fatigue. The follow-up examinations shall take place at each follow up visit , measuring those parameters recorded at the baseline examination. The further follow-up examinations shall correspond to those carried out as standard after-care investigations.

The secondary endpoints such as fatigue and quality of life shall be recorded using validated questionnaires (EORTC QLQ FA13 and EORTC QLQ BM22. All patients will also be asked to record their pain history using a pain diary (documentation of medication daily during treatment, once weekly after the end of treatment, VAS pain scale). Furthermore, the local control was assessed by means of CT images taken prior to, three and six months after RT. The pain response was documented on the VAS (range 0-10). Complete response (CR) was defined as VAS = 0 after three and six months, partial response (PR) as an improvement by at least two score points after three and six months. Overall survival (OS) was defined as time from initial diagnosis until death, bone survival as time from initial diagnosis of spinal bone metastasis until death.

In each case, the treatment plan was designed based on tumor geometry, proximity to the spinal cord, and location. The planning tumor volume (PTV) was defined as equal to gross tumor volume (GTV). The spinal cord, cauda equina, nerve roots, and bowel were contoured as organs at risk (OARs) and critical structures. An inverse treatment planning method along with a linear optimization algorithm were employed. The target volume was designated to include either the GTV and the entire vertebral body (WB group) or only the GTV (PB group) at each spinal level.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed tumor diagnosis, with secondary -diagnosed solitary/multiple spinal bone metastases
* Indication for RT of the spinal bone metastases
* Maximal two irradiated vertebral-bodies per region
* Maximal two different vertebral regions
* Age: between 18 and 80 years
* Karnofsky index (10) ≥ 70
* Signed Declaration of Informed Consent
* Tumor distance > 3 mm to myelon

Exclusion Criteria:

* Multiple myeloma or lymphoma
* Significant neurological or psychiatric disorders, including dementia and epileptic seizures
* Earlier RT at the current irradiated site
* Other severe disorders that in the judgement of the study director may prevent the patient's participation in the study
* Lacking or diminished legal capacity
* Any medical of psychological condition that the study director considers a preventive factor for the patient's ability to complete the study or to adequately
* understand the scope of the study and to give his/her consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
the time to pain relief | 3 months after treatment

SECONDARY OUTCOMES:
quality of life measured on an EORTC BM22 questionnaire | 3 and 6 months after therapy completed
Overall survival | 1 year
local control | 3 months after therapy completed
  local control as bone density is assessed 12 weeks post completion of radiotherapy using follow-up CT scan of the spine

IPD SHARING:
Plan to Share IPD: No